CLINICAL TRIAL: NCT01530659
Title: Photoreceptor Structure in A Phase 2 Study of Encapsulated Human NTC-201 Cell Implants Releasing Ciliary Neurotrophic Factor (CNTF) for Participants With Retinitis Pigmentosa Using Rates of Change in Cone Spacing and Density
Brief Title: Retinal Imaging in CNTF -Releasing Encapsulated Cell Implant Treated Patients for Early-stage Retinitis Pigmentosa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurotech Pharmaceuticals (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AOSLO-CNTF-FFB-01; FD-R-004100-01A1 (Other Grant/Funding Number: FDA OOPD)
Record Dates: First submitted 2012-01-19; First posted 2012-02-10 (Estimated); Results first posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Retinitis Pigmentosa; Usher Syndrome Type 2; Usher Syndrome Type 3
Keywords: Retinitis pigmentosa; Usher syndrome type 2; Usher syndrome type 3; Cone photoreceptor; Vision; Blind
MeSH Terms: conditions — Retinitis Pigmentosa; Usher Syndromes | interventions — Ciliary Neurotrophic Factor; Electroconvulsive Therapy; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Participants are considered in screening upon signing of the consent. Enrollment does not occur until participant is deemed eligible, as per screening, and randomized for implant. As such, there were 22 total participants enrolled in the study. There was a participant who died prior to screening procedures being conducted of which was captured in the AE section as the death occurred after consent to enter screening period. However, this participant was not enrolled as they had not completed screening or randomization for implant.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NT-501 (Experimental): Encapsulated cell therapy that delivers ciliary neurotrophic factor to the retina
  Interventions: Drug: NT-501
- Sham (Sham Comparator): Sham surgery
  Interventions: Procedure: Sham

INTERVENTIONS:
Drug: NT-501 — Study participants will undergo surgery to have an NT-501 Encapsulated Cell Therapy implant placed into the study eye.
  Other Names: CNTF, Encapsulated Cell Therapy, ECT
  Arms: NT-501
Procedure: Sham — Non-penetrating sham procedure to mimic implant procedure in the other eye.
  Arms: Sham

SUMMARY:
This clinical trial is a single-site, 30 patient study for participants who have early stage retinitis pigmentosa, or Usher syndrome (type 2 or 3). Funding Source - FDA OOPD and Foundation Fighting Blindness.

DETAILED DESCRIPTION:
This clinical trial is a prospective, randomized, double-masked, sham-controlled trial of 30 study participants who have early-stage retinitis pigmentosa, or Usher syndrome (type 2 or 3). The trial will be conducted at the University of California, San Francisco. Individuals with these diseases experience gradually worsening vision that ultimately may lead to blindness due to a genetic condition in which specialized cells in the eye's retina called photoreceptor cells cease functioning and/or die. The study is intended to use a relatively new, non-invasive technology called AOSLO (adaptive optics scanning laser ophthalmoscopy) in combination with a routine standard of care measurement called sdOCT (Spectral Domain Optical Coherence Tomography) to demonstrate that when a device that secretes an investigational drug called CNTF (Ciliary Neurotrophic Factor) is surgically placed in the patient's eye, one type of photoreceptor called "cone photoreceptors" is preserved such that the gradual loss of vision is halted.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be between 18 and 55 years of age.
2. Participant must have a diagnosis of retinitis pigmentosa or Usher Syndrome type 2 or 3 (without profound deafness or cochlear implants).
3. Participant must understand and sign the protocol informed consent. If the participant's vision is impaired to the point where he/she cannot read the informed consent document, the document will be read to the participant in its entirety.
4. Best-corrected visual acuity must be no worse than 20/63 (at least 59 letters).
5. Participants must have clear natural lenses.
6. Participants must have less than 6 diopters myopia.
7. Participants must be medically able to undergo ophthalmic surgery for the NT-501 device insertion and able to undergo all assessments and tests associated with the protocol.
8. Females of childbearing potential (women with last menses <1 year prior to screening) must agree to use an effective form of birth control from study onset until they complete the study.
9. Participants must have reproducible baseline AOSLO image at 2 baseline imaging sessions with quality suitable to identify a minimum of 7 regions of interest (ROIs) at which reliable cone spacing and/or density measures can be made over the central 5.7 degrees.
10. Participants must have interocular symmetry of disease severity as measured by cone spacing, with a difference of less than 2 standard deviations in average cone spacing z-scores at the selected ROIs between the 2 eyes.
11. Participant's clinical diagnosis must be consistent with retinal degeneration in the set of retinitis pigmentosa (RP) dystrophies.

Exclusion Criteria:

1. Participant is medically unable to comply with study procedures or follow-up visits.
2. Participant who has any of the following lens opacities: cortical opacity > standard 3, posterior subcapsular opacity > standard 3, or a nuclear opacity > standard 3 as measured on the AREDS clinical lens grading system; or participant is pseudophakic or aphakic.
3. Participant has history of corneal opacification or lack of optical clarity.
4. Participant has undergone LASIK surgery or other refractive surgery for either eye.
5. Participant has nystagmus.
6. Participant has greater than 6 diopters myopia.
7. Participant has cystoid macular edema with cysts present within 4 degrees of the foveal center that prevent acquisition of at least 7 regions of interest with clear images of cone photoreceptors.
8. Participant has fewer than 7 regions of interest (ROIs) present on 2 baseline AOSLO image montages.
9. Participant has retinal vascular disease such as diabetic retinopathy or prior retinal vascular occlusive disease.
10. Participant has chronic requirement (e.g., ≥4 weeks at a time) for ocular medications or has disease(s) that in the judgment of the examining physician are vision threatening, toxic to the lens, retina, or optic nerve or may affect the primary outcome.
11. Participant has a requirement of acyclovir and/or related products during study duration. To be eligible for this study, the participant must discontinue use of these products prior to enrollment and must not continue with the products until after they have completed the study.
12. Participant is receiving systemic steroids or other immunosuppressive medications.
13. Participant is currently participating in or has participated in any other clinical trial of a drug by ocular or systemic administration within the last 6 months.
14. Participant has previous exposure to an intra-ocular device or implant into the eye (excluding intra-ocular lens).
15. Participant has uveitis or other retinal inflammatory disease.
16. Participant has a history of myocardial infarction within the last 12 months.
17. Participant is pregnant or lactating.
18. Participant is considered immunodeficient or has a known history of HIV. A laboratory test for HIV will be performed, and a positive result is also an exclusion criterion.
19. Participant with a history of ocular herpes zoster.
20. Participant is on chemotherapy.
21. Participant has a history of malignancy, except study participant with cancer treated successfully ≥5 years prior to inclusion in the trial.
22. Participant with severe hearing disabilities in both ears.
23. Participant who has been diagnosed and treated for amblyopia as an infant.
24. Participant who, in the opinion of the study doctor, will not be a good study subject.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2012-01; Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacque Duncan, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Duncan JL, Zhang Y, Gandhi J, Nakanishi C, Othman M, Branham KE, Swaroop A, Roorda A. High-resolution imaging with adaptive optics in patients with inherited retinal degeneration. Invest Ophthalmol Vis Sci. 2007 Jul;48(7):3283-91. doi: 10.1167/iovs.06-1422. PMID 17591900
- [Background] Sieving PA, Caruso RC, Tao W, Coleman HR, Thompson DJ, Fullmer KR, Bush RA. Ciliary neurotrophic factor (CNTF) for human retinal degeneration: phase I trial of CNTF delivered by encapsulated cell intraocular implants. Proc Natl Acad Sci U S A. 2006 Mar 7;103(10):3896-901. doi: 10.1073/pnas.0600236103. Epub 2006 Feb 27. PMID 16505355
- [Background] Talcott KE, Ratnam K, Sundquist SM, Lucero AS, Lujan BJ, Tao W, Porco TC, Roorda A, Duncan JL. Longitudinal study of cone photoreceptors during retinal degeneration and in response to ciliary neurotrophic factor treatment. Invest Ophthalmol Vis Sci. 2011 Apr 6;52(5):2219-26. doi: 10.1167/iovs.10-6479. PMID 21087953

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible subjects were >18 years old with retinitis pigmentosa or Usher syndrome and adaptive optics scanning laser ophthalmoscopy (AOSLO) images in each eye with at least 7 regions having at least 50 contiguous unambiguous cones in the central 5.7 degrees of the macula at 2 baseline visits. Exclusion criteria included visual acuity worse than 20/40, lens opacity, > -6.00 D myopia, nystagmus, cystoid macular edema, retinal vascular disease, unstable fixation, and severe hearing loss.
Units Other Than Participants: Eyes
Groups:
- NT-501 Implant: A pre-determined randomization scheme will be utilized to designate each of the patient's eyes as the primary eye (to receive the NT-501 implant) or the fellow eye (Control-to receive sham surgery). Primary eye will receive the NT-501 implant
- Sham Surgery: A pre-determined randomization scheme will be utilized to designate each of the patient's eyes as the primary eye (to receive the NT-501 implant) or the fellow eye (Control-to receive sham surgery).
Period: Overall Study
Arm/Group | NT-501 Implant | Sham Surgery
Started (22 total participants and 44 eyes) | 22; 22 Eyes | 22; 22 Eyes
Completed | 22; 22 Eyes | 22; 22 Eyes
Not Completed | 0; 0 Eyes | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Population: 44 eyes of 22 patients were randomized to receive either NT-501 implant or sham surgery.
Units Other Than Participants: Eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | NT-501 Implant | Sham Surgery | Total
Number analyzed (Participants) | 22 | 22 | 22
Number analyzed (Eyes) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.8 (11.9) | 39.8 (11.9) | 39.8 (11.9)
Sex: Female, Male [Count of Units; unit: Eyes]
  Female | 9 | 9 | 18
  Male | 13 | 13 | 26
Ethnicity (NIH/OMB) [Count of Units; unit: Eyes]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 20 | 20 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Units; unit: Eyes]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 0 | 0 | 0
  White | 18 | 18 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: Eyes]
  United States | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Cone Spacing in Arcminutes (Z Score) of 2 Baseline Values Were Compared With Measurements Obtained at Post-op Month 36
Description: Average of cone spacing (nearest neighbor distance) at all regions of interest with at least 50 contiguous unambiguous cones identified over the central 5.7 degrees of the macula using confocal AOSLO at two baseline visits within each eye. Cone spacing measures were converted to Z scores based on normal mean values at similar distances from the fovea from a database of 27 age-similar normal eyes. The mean of 2 baseline cone spacing Z-score values were subtracted from the cone spacing Z score values obtained at post-op month 36
  A Z-score of 0 represents the mean cone spacing value at the distance from the fovea measured from 27 healthy subjects.
  A Z-score greater than +2 represents an abnormally increased cone spacing value at the distance from the fovea where the measurement was performed. This suggests fewer cones are present than normal at that location.
Time Frame: Post-op Month 36
Population: Measure type: difference from mean baseline to 36 months in change between intervention and control eyes in mean cone spacing Z score averaged over regions of interest in each eye.
Measure: Mean (Standard Deviation); unit: Difference in change in Z score
Units Other Than Participants: Eyes
Arm/Group | NT-501 Implant | Sham Surgery
Number analyzed (Participants) | 22 | 22
Number analyzed (Eyes) | 22 | 22
Difference in change in Z score | 1.13 (1.03) | 0.85 (1.78)

2. Secondary Outcome: Difference in logMAR Visual Acuity Change Between CNTF- and Sham Treated Eyes
Description: Difference in change in logMAR visual acuity between NT-501 and contralateral sham-treated eyes.
  Change in visual acuity was measured based on the number of letters read on a vision chart using a standard protocol. The log of the mean angle of resolution (logMAR) was used to describe the size of the smallest letters that the patient could read. A logMAR value of 0.00 corresponds to visual acuity of 20/20, a logMAR value of 0.3 corresponds to visual acuity of 20/40, a logMAR value of 0.7 corresponds to visual acuity of 20/100, and a logMAR value of 1.00 corresponds to visual acuity of 20/200.
Time Frame: Post-op Month 36
Population: Difference in change in logMAR visual acuity between NT-501 and contralateral sham-treated eyes.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | NT-501 Implant | Sham Surgery
Number analyzed (Participants) | 22 | 22
Number analyzed (Eyes) | 22 | 22
logMAR | 0.004 (0.010) | 0.014 (0.082)

ADVERSE EVENTS:
Time Frame: Serious and Other (Not Including Serious) Adverse Events were collected only for randomized participants through study completion, an average of 36 months. However, mortality is noted for one participant who passed away due to unrelated issues before being randomized.
Description: Non-ocular, Non-serious adverse events were not required to be collected per protocol. All-Cause Mortality and Non-Ocular Serious Adverse Events are reported at the participant level. Ocular Serious and Other (Not Including Serious) Adverse Events are presented with total number of eyes monitored/assessed as the at Risk population.
Groups:
- Prior to Randomization: One participant was consented and enrolled but died before being randomized to receive the study intervention.
Arm/Group | NT-501 Implant | Sham Surgery | Prior to Randomization
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22 | 1/1
Serious Adverse Events (participants affected / at risk) | 4/22 | 4/22 | 0/0
Other Adverse Events (participants affected / at risk) | 2/22 | 1/22 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NT-501 Implant (N=22) | Sham Surgery (N=22) | Prior to Randomization (N=0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0 (0)
Reversible Cardiac Vasospasm (Cardiac disorders) | 1 | 1 | 0 (0)
Total Eye Disorders (Eye disorders) | 4 (5) | 1 (1) | 0 (0)
Clinically Significant Cystoid Macular Edema (Eye disorders) | 1 | 0 | 0 (0)
Secondary Surgical Intervention (excluding Posterior Capsulotomy) (Eye disorders) | 1 | 1 | 0 (0) — Bilateral cataract extraction at 30 months required early NT-501 implant removal.
Ocular discomfort (Eye disorders) | 1 | 0 | 0 (0)
Reduced peripheral visual field (Eye disorders) | 1 | 0 | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NT-501 Implant (N=22) | Sham Surgery (N=22) | Prior to Randomization (N=0)
Epiretinal membrane (Eye disorders) | 1 | 0 | NA
Pelvic fracture (Musculoskeletal and connective tissue disorders) | 1 | 1 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2015-10-27): https://cdn.clinicaltrials.gov/large-docs/59/NCT01530659/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-20): https://cdn.clinicaltrials.gov/large-docs/59/NCT01530659/SAP_001.pdf